CLINICAL TRIAL: NCT03175354
Title: A Multicenter, Randomized, Double-Blind, Bilateral, Vehicle-Controlled Study of the Safety and Efficacy of ALX-101 Topical Gel Administered Twice Daily in Adult and Adolescent Subjects With Moderate Atopic Dermatitis
Brief Title: A Study in Subjects With Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ralexar Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALX-101-ATOP-202
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Atopic Dermatitis; Eczema, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALX-101 Gel 1.5% vs. ALX-101 Gel Vehicle (Experimental): ALX-101 Gel 1.5% applied twice daily for 42 days to one treatment area and ALX-101 Gel Vehicle applied twice daily for 42 days to a second treatment area. Treatments will be randomly assigned to bilateral target areas.
  Interventions: Drug: ALX-101 Gel 1.5% and ALX-101 Gel Vehicle
- ALX-101 Gel 5% vs. ALX-101 Gel Vehicle (Experimental): ALX-101 Gel 5% applied twice daily for 42 days to one treatment area and ALX-101 Gel Vehicle applied twice daily for 42 days to a second treatment area. Treatments will be randomly assigned to bilateral target areas.
  Interventions: Drug: ALX-101 Gel 5% and ALX-101 Gel Vehicle

INTERVENTIONS:
Drug: ALX-101 Gel 1.5% and ALX-101 Gel Vehicle — Bilateral application of ALX-101 Gel 1.5% and ALX-101 Gel Vehicle
  Arms: ALX-101 Gel 1.5% vs. ALX-101 Gel Vehicle
Drug: ALX-101 Gel 5% and ALX-101 Gel Vehicle — Bilateral application of ALX-101 Gel 5% and ALX-101 Gel Vehicle
  Arms: ALX-101 Gel 5% vs. ALX-101 Gel Vehicle

SUMMARY:
This is a randomized, double-blind, vehicle-controlled study to evaluate the safety and efficacy of ALX-101 Gel 1.5% and 5% and a matching ALX-101 Gel Vehicle when applied topically twice daily for 42 days to adult and adolescent subjects with moderate atopic dermatitis.

DETAILED DESCRIPTION:
The main objectives of this study are to:

* Evaluate the safety and tolerability of ALX-101 Gel 1.5% and 5% when applied topically in subjects with moderate atopic dermatitis compared with a matching ALX-101 Gel Vehicle
* Evaluate the dose-response relationship of ALX-101 Gel 1.5% and 5% when applied topically twice daily in subjects with moderate atopic dermatitis compared with a matching ALX-101 Gel Vehicle.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for the study, subjects must fulfill all of the following criteria:

1. Subject is at least 12 years of age
2. Subject has a clinical diagnosis of stable AD characterized by:

   1. Pruritus
   2. Eczema (acute, subacute, chronic)

      * Typical morphology and distribution with age-specific patterns
      * Chronic or relapsing history
3. Subject must have active AD covering 4-24% body surface area (BSA) (right and left treatment areas combined)
4. Bilateral treatment areas of AD must be 5 cm apart
5. Presence of AD with comparable bilateral target evaluation areas on (right and left sides of body) and within each bilateral treatment area:

   a. Bilateral target evaluation areas must each have active AD covering 0.5 -2% body surface area (BSA)
6. Bilateral target evaluation areas of AD must each have a Physician's Global Assessment score of 3 ("moderate") to be treated
7. Subject Visit 1 photographs are approved for enrollment by dermatology assessor
8. If the subject is a woman of childbearing potential, she has a negative urine pregnancy test and agrees to use an approved effective method of birth control for the duration of the study
9. Subject is non-pregnant and non-lactating
10. Subject is in good general health and free of any known disease state or physical condition which, in the investigator's opinion, might impair evaluation of the AD being treated or which exposes the subject to an unacceptable risk by study participation
11. Subject is willing and able to follow all study instructions and to attend all study visits
12. Subject is able to comprehend and willing to sign an Informed Consent Form (ICF)/Assent Form (AF)
13. Parent/guardian has the ability to understand, agree to and sign the study Informed Consent Form (ICF) prior to initiation of any protocol-related procedures as applicable; subject has the ability to give assent in the Assent Form (AF)
14. All female subjects of childbearing potential must use acceptable methods of contraception from the Screening Visit continuously until 14 days after stopping study drug.

Exclusion Criteria:

Any subject who meets one or more of the following criteria will not be included in this study:

1. Subject has spontaneously improving or rapidly deteriorating AD
2. Subject has clinically infected AD
3. Subject has any signs or symptoms associated with topical AD therapy (e.g., history of anaphylaxis, hypersensitivity reactions, skin atrophy, striae, pigmentary changes) which, in the investigator's opinion, might impair evaluation of the AD being treated or which exposes the subject to an unacceptable risk by study participation
4. Subject has used any systemic immunosuppressive or immunomodulatory therapy (e.g., etanercept, alefacept, infliximab) within 16 weeks prior to Visit 1
5. Subject has used any phototherapy (e.g., ultraviolet A, ultraviolet B) which, in the investigator's opinion, might affect AD within 4 weeks prior to Visit 1
6. Subject has used any systemic therapy (e.g., systemic corticosteroids [intranasal and inhaled corticosteroids are allowed]), prednisone cyclosporine, immunosuppressants/immunomodulators, Janus Kinase (JAK) inhibitors, methotrexate, cytostatics) within 4 weeks prior to Visit 1 which, in the investigator's opinion, might impair evaluation of the AD being treated or which exposes the subject to an unacceptable risk by study participation
7. Subject has used any systemic antibiotics within 2 weeks prior to Visit 1
8. Subject has used any topical AD therapy (e.g., corticosteroids, calcineurin inhibitors, topical H1 and H2 antihistamines, topical antimicrobials, and other medicated topical agents) on the planned treatment area(s) within one week prior to Visit 1
9. Subject has used emollients/moisturizers on the planned treatment area(s) within 4 hours prior to Visit 1
10. Subject is currently using H1 antihistamines (e.g., diphenhydramine, terfenadine) UNLESS a stable dose has been used for at least 14 days prior to Visit 1
11. Subject has a history of sensitivity to any of the ingredients in the study medications
12. Subject has any known concomitant dermatologic or medical condition which, in the investigator's opinion, might impair evaluation of the bilateral treatment and/or target evaluation areas of AD being treated or which exposes the subject to an unacceptable risk by study participation (e.g., psoriasis, lichen planus, lichen simplex chronicus,…)
13. Subject has participated in an investigational drug trial in which administration of an investigational study medication occurred within 30 days prior to Visit 1.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Physician's Global Assessment (PGA) | Day 42
  The primary effectiveness analysis will be based on mean change in PGA score from baseline (Visit 2) to Visit 6.

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Ralexar Investigational Site 35, Anniston, Alabama
  - Ralexar Investigational Site 21, Birmingham, Alabama
  - Ralexar Investigational Site 18, Laguna Hills, California
  - Ralexar Investigational Site 23, Los Angeles, California
  - Ralexar Investigational Site 24, Oceanside, California
  - Ralexar Investigational Site 34, San Diego, California
  - Ralexar Investigational Site 16, San Diego, California
  - Ralexar Investigational Site 33, San Diego, California
  - Ralexar Investigational Site 27, Santa Monica, California
  - Ralexar Investigational Site 1, Miami, Florida
  - Ralexar Investigational Site 14, Pinellas Park, Florida
  - Ralexar Investigational Site 22, Tampa, Florida
  - Ralexar Investigational Site 29, Snellville, Georgia
  - Ralexar Investigational Site 17, New Albany, Indiana
  - Ralexar Investigational Site 32, Louisville, Kentucky
  - Ralexar Investigational Site 7, Louisville, Kentucky
  - Ralexar Investigational Site 11, Warren, Michigan
  - Ralexar Investigational Site 15, Fridley, Minnesota
  - Ralexar Investigational Site 25, Saint Joseph, Missouri
  - Ralexar Investigational Site 26, Albuquerque, New Mexico
  - Ralexar Investigational Site 20, New York, New York
  - Ralexar Investigational Site 30, Stony Brook, New York
  - Ralexar Investigational Site 28, Charlotte, North Carolina
  - Ralexar Investigational Site 12, Beachwood, Ohio
  - Ralexar Investigational Site 5, Cincinnati, Ohio
  - Ralexar Investigational Site 3, Oklahoma City, Oklahoma
  - Ralexar Investigational Site 8, Johnston, Rhode Island
  - Ralexar Investigational Site 6, Spartanburg, South Carolina
  - Ralexar Investigational Site 9, Nashville, Tennessee
  - Ralexar Investigational Site 19, Austin, Texas
  - Ralexar Investigational Site 31, Austin, Texas
  - Ralexar Investigational Site 4, Plano, Texas
  - Ralexar Investigational Site 2, San Antonio, Texas
  - Ralexar Investigational Site 13, Richmond, Virginia
  - Ralexar Investigational Site 10, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Undecided